CLINICAL TRIAL: NCT06763497
Title: The Efficacy of Systematic Oral Feeding Education Program (SOFEP) on Feeding Techniques, Caregiver Stress, and Infant Feeding Skills in Caregivers of Infants With Congenital Heart Disease After Surgery
Brief Title: The Efficacy of Systematic Oral Feeding Education Program
Acronym: SOFEP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, National Taiwan University Clinical Trial Center, Nurse, National Taiwan University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 202412004RINA
Record Dates: First submitted 2025-01-01; First posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2024-12

CONDITIONS: Congenital Heart Disease
Keywords: Congenital Heart Disease; Oral Feeding; Systematic Health Education Program; Feeding Difficulties; Parenting Stress
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The control group - received routine care (No Intervention): On the day of receipt of the case, after completing the informed consent form, the pre-test was also completed, including asking the subjects to complete the "Basic Case Information Form" and the "Parenting Stress Scale", and the researcher observed the primary caregiver feeding the baby. , use the "Oral Feeding Techniques Scale" to evaluate the caregiver's feeding techniques and the "Infant Feeding Skills Assessment Scale" to evaluate the infant's oral feeding status. In addition, the subjects were asked to fill in the feeding record form every day during the 14-day period, and complete the aforementioned self-report scale and observation evaluation form on the day the case was closed. The control group received routine care in the ward and took the post-test of the scale on the 14th day.
- experimental group - systematic oral feeding education program (Other): The experimental group conducted 11 interventions before and after completing the primary caregiver's oral feeding techniques, caregiving stress and infant feeding skills. The first time was after completing the pre-test, a systematic oral feeding education program was used to provide feeding skills guidance and Practical feeding guidance, and assisting in video recording during the actual feeding operation. After completion, the video was used to discuss possible corrections. The remaining 10 interventions were conducted on days 2-4, 6-9, and 11-13 to observe the main care every day. The patient's feeding status was reviewed once and assistance and suggestions were provided. On the 14th day, the patient completed the relevant scale post-test.
  Interventions: Other: Systematic Oral Feeding Education Program

INTERVENTIONS:
Other: Systematic Oral Feeding Education Program — The experimental group will receive 11 intervention sessions during the study period. The first intervention will occur immediately after the pretest and will involve a systematic oral feeding education program, including guided feeding techniques and practical feeding demonstrations. During the feeding session, caregivers' practices will be recorded on video. These recordings will then be reviewed with the caregiver to identify areas for improvement.The remaining 10 intervention sessions will take place daily on days 2-4, 6-9, and 11-13, during which the researcher will observe the primary caregiver's feeding practices, provide assistance, and offer tailored suggestions. On the 14th day, the experimental group will complete the same posttest assessments as the control group.
  Arms: experimental group - systematic oral feeding education program

SUMMARY:
After the intervention of Systematic Oral Feeding Education Program:

1. The feeding techniques scores of the main caregivers in the experimental group will be higher than those in the control group.
2. The caregiving stress scores of the main caregivers in the experimental group will be lower than those in the control group.
3. The feeding skill scores of infants in the experimental group will be higher than those in the control group.

DETAILED DESCRIPTION:
This study will adopt a quasi-experimental design and will purposively and consecutively sample participants from the pediatric ward of a medical center in northern Taiwan. Enrollment will be conducted based on the inclusion and exclusion criteria of the study. To avoid contamination between the experimental and control groups, recruitment for the control group will be completed before recruitment for the experimental group begins. Each group will undergo a 3-month recruitment period or until 30 participants have been enrolled in each group.

Each participant will be followed for 14 days. On the enrollment day, after obtaining informed consent, a pretest will be conducted. This includes completing the "Participant Demographic Information Form" and the "Parenting Stress Index" and having the primary caregiver's infant feeding practices observed by the researcher. The caregiver's feeding techniques will be assessed using the "Oral Feeding Techniques Scale," and the infant's oral feeding performance will be evaluated using the "Early Feeding Skills Assessment Scale." Additionally, participants will complete a daily feeding log for the 14-day study period. On the final day, posttests will include the same self-reported questionnaires and observation-based assessments as the pretest.

The control group will receive standard ward care and will complete the posttest on the 14th day. The experimental group will receive 11 intervention sessions during the study period. The first intervention will occur immediately after the pretest and will involve a systematic oral feeding education program, including guided feeding techniques and practical feeding demonstrations. During the feeding session, caregivers' practices will be recorded on video. These recordings will then be reviewed with the caregiver to identify areas for improvement.

The remaining 10 intervention sessions will take place daily on days 2-4, 6-9, and 11-13, during which the researcher will observe the primary caregiver's feeding practices, provide assistance, and offer tailored suggestions. On the 14th day, the experimental group will complete the same posttest assessments as the control group.

Statistical analysis will be conducted using SPSS Statistics (version 22.0). Independent sample t-tests, paired sample t-tests, and generalized estimating equations (GEE) will be employed to evaluate the effects of the systematic oral feeding education program on the primary caregiver's feeding techniques, caregiving stress, and the infant's oral feeding skills.

ELIGIBILITY:
Infants with congenital heart disease and their primary caregivers who meet the following conditions will be admitted:

1. Infant Criteria:

   Inclusion Criteria:
   * Infants diagnosed with congenital heart disease and younger than 12 months at the time of enrollment.
   * Infants unable to meet their required oral feeding volume (10% of body weight = 100 ml/kg) at the time caregiving begins.
   * Infants who have undergone open-heart surgery with cardiopulmonary bypass.
   * Infants assessed by physicians as ready to begin oral feeding training.

   Exclusion Criteria:
   * Corrected gestational age less than 32 weeks.
   * Infants with congenital conditions involving the mouth, throat, or esophagus (e.g., cleft palate, esophageal atresia with tracheoesophageal fistula).
   * Infants with congenital central nervous system disorders.
   * Infants consuming food via methods other than bottle feeding (e.g., spoon-feeding, complementary food, or solid food).
   * Infants whose primary feeding method is breastfeeding directly at the breast.
2. Primary Caregiver Criteria

Inclusion Criteria:

* Caregivers aged 18 years or older.
* The infant's legal father or mother.
* Caregivers who participate in at least two oral feeding sessions per day for the infant.

Exclusion Criteria:

* Caregivers unable to complete self-administered questionnaires.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-12-19 (Estimated); Study Completion 2025-12-19 (Estimated)

PRIMARY OUTCOMES:
oral feeding techniques scale for primary caregivers early feeding skills assessment EFS parenting stress index, fourth edition short form, PSI-4-SF | on the 14th day
  The researcher developed a self-designed scale based on systematic oral feeding education program, expert opinions, and relevant literature to evaluate the primary caregiver's oral feeding techniques. The scale comprises four main sections:
  1. Preparation before feeding (including oral stimulation).
  2. Feeding process (including oral support).
  3. Provision of developmental feeding support.
  4. Observation of dehydration warning signs. The scale consists of 21 items. When the caregiver's feeding behavior or response aligns with the descriptions in the items, it is marked as "Yes" and awarded 1 point. If not, it is marked as "No" and receives 0 points. The total score ranges from 0 to 21, with higher scores indicating better feeding techniques.
  The evaluation is conducted by observing the caregiver during actual feeding sessions (or reviewing recorded feeding videos) and scoring based on their observed behaviors.
early feeding skills assessment, EFS | on the 14th day
  The EFS consists of 24 items that assess infant feeding skills across three domains:
  1. Preparation for oral feeding (3 items: motor behavior, state, and oral behaviors when given a pacifier).
  2. Feeding process evaluation, which des: breathing regulation (5 items), coordination of oral movements (4 items), swallowing coordination (4 items), sustaining engagement (2 items), and physiological stability (4 items).
  3. Post-feeding tolerance (2 items: state and energy level). Each item is scored on a scale of 1 to 3, where a score of 1 indicates problems, and a score of 3 indicates no problems. The total score ranges from 24 to 72, with higher scores indicating better feeding skills.
  The assessment identifies both the infant's abilities and areas of difficulty.
parenting stress index, fourth edition short form, PSI-4-SF | on the 14th day
  This scale was originally developed to evaluate parenting stress in parents of children. Parenting Stress Index, Fourth Edition Short Form (PSI-4-SF) consists of 36 items selected from the Long Form and is divided into three subscales:
  1. Parental Distress (Items 1-12): Assesses the distress experienced by individuals in their role as a parent.
  2. Parent-Child Dysfunctional Interaction (Items 13-24): Evaluates stress arising from interactions and mutual influences between parents and children.
  3. Difficult Child (Items 25-36): Assesses behavioral characteristics of the child that contribute to stress in the parent-child system.
  The scale uses a 5-point Likert scale for scoring, ranging from 1 ("Strongly Disagree") to 5 ("Strongly Agree"). The total score ranges from a minimum of 36 to a maximum of 180, with higher scores indicating greater levels of parenting stress.

CONTACTS AND LOCATIONS:
Overall Officials: YA-HAN LIN, MS, Principal Investigator

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bala P, Kaur R, Mukhopadhyay K, Kaur S. Oromotor Stimulation for Transition from Gavage to Full Oral Feeding in Preterm Neonates: A Randomized controlled trial. Indian Pediatr. 2016 Jan;53(1):36-8. doi: 10.1007/s13312-016-0786-3. PMID 26840669
- [Background] Desai, H., & Lim, A. N. (2019). Neurodevelopmental intervention strategies to improve oral feeding skills in infants with congenital heart defects. Perspectives of the ASHA Special Interest Groups, 4(6), 1492-1497.
- [Background] Desai H, Jones CE, Fogel JL, Negrin KA, Slater NL, Morris K, Doody LR, Engstler K, Torzone A, Smith J, Butler SC. Assessment and management of feeding difficulties for infants with complex CHD. Cardiol Young. 2023 Jan;33(1):1-10. doi: 10.1017/S1047951122004024. Epub 2022 Dec 23. PMID 36562257
- [Background] Fucile S, Dow K. A Unique Clinical Tool for the Evaluation of Oral Feeding Skills in Infants. Can J Occup Ther. 2023 Sep;90(3):240-248. doi: 10.1177/00084174221134738. Epub 2022 Oct 30. PMID 36314405
- [Background] Fucile S, Gisel E, Lau C. Oral stimulation accelerates the transition from tube to oral feeding in preterm infants. J Pediatr. 2002 Aug;141(2):230-6. doi: 10.1067/mpd.2002.125731. PMID 12183719
- [Background] Goday PS, Huh SY, Silverman A, Lukens CT, Dodrill P, Cohen SS, Delaney AL, Feuling MB, Noel RJ, Gisel E, Kenzer A, Kessler DB, Kraus de Camargo O, Browne J, Phalen JA. Pediatric Feeding Disorder: Consensus Definition and Conceptual Framework. J Pediatr Gastroenterol Nutr. 2019 Jan;68(1):124-129. doi: 10.1097/MPG.0000000000002188. PMID 30358739
- [Background] Goldstein SA, Watkins KJ, Lowery RE, Yu S, Knight RM, Drayton AK, Sayers L, Gaies M. Oral Aversion in Infants With Congenital Heart Disease: A Single-Center Retrospective Cohort Study. Pediatr Crit Care Med. 2022 Mar 1;23(3):e171-e179. doi: 10.1097/PCC.0000000000002879. PMID 34991136
- [Background] Greene Z, O'Donnell CP, Walshe M. Oral stimulation for promoting oral feeding in preterm infants. Cochrane Database Syst Rev. 2016 Sep 20;9(9):CD009720. doi: 10.1002/14651858.CD009720.pub2. PMID 27644167
- [Background] Hasenstab KA, Jadcherla SR. Evidence-Based Approaches to Successful Oral Feeding in Infants with Feeding Difficulties. Clin Perinatol. 2022 Jun;49(2):503-520. doi: 10.1016/j.clp.2022.02.004. PMID 35659100
- [Background] Hewitt-Taylor J. Clinical guidelines and care protocols. Intensive Crit Care Nurs. 2004 Feb;20(1):45-52. doi: 10.1016/j.iccn.2003.08.002. PMID 14726253
- [Background] Holst LM, Serrano F, Shekerdemian L, Ravn HB, Guffey D, Ghanayem NS, Monteiro S. Impact of feeding mode on neurodevelopmental outcome in infants and children with congenital heart disease. Congenit Heart Dis. 2019 Nov;14(6):1207-1213. doi: 10.1111/chd.12827. Epub 2019 Aug 2. PMID 31373176
- [Background] Horsley M, Hill GD, Kaskie S, Schnautz M, Brown J, Marcuccio E. Evaluation of an Outpatient and Telehealth Initiative to Reduce Tube Dependency in Infants with Complex Congenital Heart Disease. Pediatr Cardiol. 2022 Oct;43(7):1429-1437. doi: 10.1007/s00246-022-02864-6. Epub 2022 Mar 25. PMID 35333946
- [Background] Indramohan G, Pedigo TP, Rostoker N, Cambare M, Grogan T, Federman MD. Identification of Risk Factors for Poor Feeding in Infants with Congenital Heart Disease and a Novel Approach to Improve Oral Feeding. J Pediatr Nurs. 2017 Jul-Aug;35:149-154. doi: 10.1016/j.pedn.2017.01.009. Epub 2017 Feb 4. PMID 28169036
- [Background] Jones CE, Desai H, Fogel JL, Negrin KA, Torzone A, Willette S, Fridgen JL, Doody LR, Morris K, Engstler K, Slater NL, Medoff-Cooper B, Smith J, Harris BD, Butler SC. Disruptions in the development of feeding for infants with congenital heart disease. Cardiol Young. 2021 Apr;31(4):589-596. doi: 10.1017/S1047951120004382. Epub 2020 Dec 11. PMID 33303052
- [Background] Jones C, Winder M, Ou Z, Miller TA, Malik L, Flannery M, Glotzbach K. Feeding outcomes in post-discharge feeding clinic for infants following cardiac surgery. Cardiol Young. 2022 Apr;32(4):628-635. doi: 10.1017/S1047951121002833. Epub 2021 Jul 26. PMID 34304751
- [Background] Kamran, F., Sagheb, S., Khatoonabadi, S. A., Ebadi, A., Faryadras, Y., & Aghajanzadeh, M. (2021). The Validity and Reliability of Early Feeding Skills Assessment and Cue-Based Feeding Scales for Preterm Infants. Middle East Journal of Rehabilitation and Health Studies, 8(3). https://doi.org/10.5812/mejrh.110973
- [Background] Kotowski J, Fowler C, Hourigan C, Orr F. Bottle-feeding an infant feeding modality: An integrative literature review. Matern Child Nutr. 2020 Apr;16(2):e12939. doi: 10.1111/mcn.12939. Epub 2020 Jan 6. PMID 31908144
- [Background] Krom H, de Winter JP, Kindermann A. Development, prevention, and treatment of feeding tube dependency. Eur J Pediatr. 2017 Jun;176(6):683-688. doi: 10.1007/s00431-017-2908-x. Epub 2017 Apr 13. PMID 28409284
- [Background] Lau C, Geddes D, Mizuno K, Schaal B. The development of oral feeding skills in infants. Int J Pediatr. 2012;2012:572341. doi: 10.1155/2012/572341. Epub 2012 Nov 5. No abstract available. PMID 23193413
- [Background] Mahoney AS, O'Donnell M, Coyle JL, Turner R, White KE, Skoretz SA. Non-Pharmacological and Non-Surgical Feeding Interventions for Hospitalized Infants with Pediatric Feeding Disorder: A Scoping Review. Dysphagia. 2023 Jun;38(3):818-836. doi: 10.1007/s00455-022-10504-7. Epub 2022 Aug 31. PMID 36044080
- [Background] Manno, C. J., Fox, C., Eicher, P. S., & Kerwin, M. E. (2005). Early oral-motor interventions for pediatric feeding problems: What, when and how. Journal of Early and Intensive Behavior Intervention, 2(3), 145. https://doi.org/10.1037/h0100310
- [Background] Martini S, Beghetti I, Annunziata M, Aceti A, Galletti S, Ragni L, Donti A, Corvaglia L. Enteral Nutrition in Term Infants with Congenital Heart Disease: Knowledge Gaps and Future Directions to Improve Clinical Practice. Nutrients. 2021 Mar 13;13(3):932. doi: 10.3390/nu13030932. PMID 33805775
- [Background] Medoff-Cooper B, Irving SY, Hanlon AL, Golfenshtein N, Radcliffe J, Stallings VA, Marino BS, Ravishankar C. The Association among Feeding Mode, Growth, and Developmental Outcomes in Infants with Complex Congenital Heart Disease at 6 and 12 Months of Age. J Pediatr. 2016 Feb;169:154-9.e1. doi: 10.1016/j.jpeds.2015.10.017. Epub 2015 Nov 13. PMID 26585995
- [Background] Morag I, Hendel Y, Karol D, Geva R, Tzipi S. Transition From Nasogastric Tube to Oral Feeding: The Role of Parental Guided Responsive Feeding. Front Pediatr. 2019 May 9;7:190. doi: 10.3389/fped.2019.00190. eCollection 2019. PMID 31143759
- [Background] Neto, F., França, A. P., & Cruz, S. (2016). An algorithm proposal to oral feeding in premature infants. The European Procedings of Social Behavioural Sciences, 87-98. https://doi.org/10.15405/epsbs.2016.07.02.8
- [Background] Philbin MK, Ross ES. The SOFFI Reference Guide: text, algorithms, and appendices: a manualized method for quality bottle-feedings. J Perinat Neonatal Nurs. 2011 Oct-Dec;25(4):360-80. doi: 10.1097/JPN.0b013e31823529da. PMID 22071621
- [Background] Ross ES, Browne JV. Developmental progression of feeding skills: an approach to supporting feeding in preterm infants. Semin Neonatol. 2002 Dec;7(6):469-75. doi: 10.1053/siny.2002.0152. PMID 12614599
- [Background] Ross ES, Philbin MK. Supporting oral feeding in fragile infants: an evidence-based method for quality bottle-feedings of preterm, ill, and fragile infants. J Perinat Neonatal Nurs. 2011 Oct-Dec;25(4):349-57; quiz 358-9. doi: 10.1097/JPN.0b013e318234ac7a. PMID 22071619
- [Background] Slater, N., Spader, M., Fridgen, J., Horsley, M., Davis, M., & Griffin, K. H. (2021). Weaning from a feeding tube in children with congenital heart disease: A review of the literature. Progress in Pediatric Cardiology, 62, 101406. https://doi.org/10.1016/j.ppedcard.2021.101406
- [Background] Thoyre SM, Hubbard C, Park J, Pridham K, McKechnie A. Implementing Co-Regulated Feeding with Mothers of Preterm Infants. MCN Am J Matern Child Nurs. 2016 Jul/Aug;41(4):204-211. doi: 10.1097/NMC.0000000000000245. PMID 27111440
- [Background] Thoyre SM, Pados BF, Shaker CS, Fuller K, Park J. Psychometric Properties of the Early Feeding Skills Assessment Tool. Adv Neonatal Care. 2018 Oct;18(5):E13-E23. doi: 10.1097/ANC.0000000000000537. PMID 30239407
- [Background] Thoyre SM, Shaker CS, Pridham KF. The early feeding skills assessment for preterm infants. Neonatal Netw. 2005 May-Jun;24(3):7-16. doi: 10.1891/0730-0832.24.3.7. PMID 15960007
- [Background] Ubeda Tikkanen A, Vova J, Holman L, Chrisman M, Clarkson K, Santiago R, Schonberger L, White K, Badaly D, Gauthier N, Pham TDN, Britt JJ, Crouter SE, Giangregorio M, Nathan M, Akamagwuna UO. Core components of a rehabilitation program in pediatric cardiac disease. Front Pediatr. 2023 May 31;11:1104794. doi: 10.3389/fped.2023.1104794. eCollection 2023. PMID 37334215
- [Background] White, A., & Parnell, K. (2013). The transition from tube to full oral feeding (breast or bottle)-A cue-based developmental approach. Journal of Neonatal Nursing, 19(4), 189-197. https://doi.org/10.1016/j.jnn.2013.03.006
- [Background] Willson, L., & Spence, K. (2022). Development of a Foundation Protocol for Feeding Complex Care Neonates and Enablers and Barriers to Its Implementation. Comprehensive Child and Adolescent Nursing, 45(3), 331-344. https://doi.org/10.1080/24694193.2022.2053613
- See also: American Heart Association. (n.d.). The Impact of Congenital Heart Defects. — https://www.heart.org/en/health-topics/congenital-heart-defects/the-impact-of-congenital-heart-defects
- See also: Thoyre, S. (2021). Early Feeding Skills Assessment Tool (EFS). Retrieved from Feeding Flock. — https://feedingflockteam.org/wp-content/uploads/2023/11/EFS-Clinical-Version-2023-8-6-1.pdf